CLINICAL TRIAL: NCT03023709
Title: Tissue-specific Responses to Influenza Immunization and Their Relation to Blood Biomarkers. U19-HIPC Vaccination and Infection: Indicators of Immunological Health and Responsiveness
Brief Title: Tissue-specific Responses to Influenza Immunization and Their Relation to Blood Biomarkers (SLVP032)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the ACIP guidelines halting the use of LAIV
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SU-33722; 2U19AI057229-11 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Quadrivalent inactivated influenza vaccine; Quadrivalent live, attenuated influenza vaccine; Adults with obstructive sleep apnea
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Intervention Model Description: 3-5 participants will receive quadrivalent inactivated flu (IIV4) vaccine as a pilot study to establish protocols for immune cell isolation. Once the pilot study ends, all new participants will receive live, attenuated influenza vaccine and IIV4 will no longer be utilitzed.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilot phase (Other): Participants will receive the current seasonal quadrivalent, inactivated influenza vaccine (IIV4)/Fluzone® given intramuscularly to confirm the safety of administering the seasonal influenza vaccine 3-14 days prior to tonsillectomy.
  Interventions: Biological: Fluzone®
- Study phase (Other): Participants will be given the current year's quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4)/FluMist® intranasally 3-14 days prior to tonsillectomy.
  Interventions: Biological: FluMist®

INTERVENTIONS:
Biological: Fluzone® — quadrivalent, inactivated influenza virus vaccine, intramuscular
  Arms: Pilot phase
Biological: FluMist® — quadrivalent, live, attenuated influenza vaccine, intranasal spray
  Arms: Study phase

SUMMARY:
The investigators collected blood and lymphoid tissues routinely discarded during surgery from adults after a routine seasonal influenza vaccination to determine how immune memory develops at the actual site of infection, and how immunization may alter this process.

DETAILED DESCRIPTION:
This is a Phase IV study of licensed influenza vaccines with up to 30 male and female adults, 18-49 years of age that was halted due to the recommendation that live, attenuated influenza vaccine (LAIV) not be used as a seasonal flu vaccine. Volunteers were patients undergoing tonsillectomy for treatment of obstructive sleep apnea (OSA).

In the initial pilot phase of the study, up to 3 volunteers will be enrolled and will receive the current seasonal quadrivalent, inactivated influenza vaccine (IIV4) given intramuscularly to confirm the safety of administering the seasonal influenza vaccine 3-14 days prior to tonsillectomy. Enrollment of the remaining study volunteers into the main portion of the study will begin once the initial pilot phase is completed. All of the remaining study volunteers will be given the current year's quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4) intranasally.

The second study visit for all volunteers will occur at the time of the volunteer's tonsillectomy surgery, 3-14 days after Visit 01. A member of the surgical team will collect a 20 mL blood sample and a sample of the resected tonsil tissue that would otherwise be discarded to be distributed to the lab.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy 18-49 year old male and female patients undergoing tonsillectomy for obstructive sleep apnea.
2. Willing to complete the informed consent process
3. Availability for follow-up for the planned duration of the study
4. Acceptable medical history by review of inclusion/exclusion criteria

Exclusion Criteria:

1. Prior off-study vaccination with seasonal influenza vaccine within three months of study vaccination
2. Life-threatening reactions to previous influenza vaccinations
3. Asthma (contraindication for receipt of LAIV4) for study volunteers; not a contraindication for enrolling as a pilot phase volunteer receiving IIV4.
4. Allergy to egg or egg products or to vaccine components (including gentamicin, gelatin, arginine or MSG for participants receiving LAIV4).
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function; may include significant liver disease, diabetes mellitus treated with insulin or moderate to severe renal disease
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C.
10. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
11. Participants who care for severely immunosuppressed persons that require a protective environment should not receive LAIV, or should avoid contact with such persons for 7 days after receipt, given the theoretical risk for transmission of the live attenuated vaccine virus to close contacts. [If yes, may be ineligible]
12. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
13. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator might jeopardize volunteer safety or compliance with the protocol.
14. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
15. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox will be reviewed by investigators to determine if study participation would affect the volunteer's safety or compliance with the protocol.
16. Has taken an influenza antiviral medication within 48 hours prior to study vaccination [For volunteers receiving LAIV; If yes, may not eligible if unable to schedule at an appropriate interval].
17. Receipt of blood or blood products within the past 6 months or planned use during the study.
18. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
19. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit (~ 14 days after study vaccination)
20. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 14 days after study enrollment)
21. Need for allergy immunization (that cannot be postponed) until after the last study visit.
22. History of Guillain-Barré syndrome
23. Pregnant woman;
24. Breastfeeding woman [if volunteer will receive LAIV4]
25. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
26. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or donation of platelets within 2 weeks of enrollment or planned donation prior to completion of the last visit.
27. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was halted after the IIV pilot phase because the LAIV vaccine for the study phase was not recommended for use by ACIP so no participants enrolled in the LAIV study phase.
Groups:
- Pilot Phase (IIV4): Participants will receive the seasonal quadrivalent, inactivated influenza vaccine (IIV4), Fluzone®, given intramuscularly to confirm the safety of administering licensed seasonal influenza vaccine 3-14 days prior to tonsillectomy.
  Fluzone®: quadrivalent, inactivated influenza virus vaccine, intramuscular
- Study Phase (LAIV4): Participants will be given the quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4), FluMist®, intranasally 3-14 days prior to tonsillectomy.
  FluMist®: quadrivalent, live, attenuated influenza vaccine, intranasal spray
Period: Overall Study
Arm/Group | Pilot Phase (IIV4) | Study Phase (LAIV4)
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot Phase (IIV4): Participants will receive the seasonal quadrivalent, inactivated influenza vaccine (IIV4), Fluzone®, given intramuscularly to confirm the safety of administering the seasonal influenza vaccine 3-14 days prior to tonsillectomy.
  Fluzone®: quadrivalent, inactivated influenza virus vaccine, intramuscular
- Study Phase (LAIV4): Participants will be given quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4), FluMist®, intranasally 3-14 days prior to tonsillectomy.
  FluMist®: quadrivalent, live, attenuated influenza vaccine, intranasal spray
- Total: Total of all reporting groups
Arm/Group | Pilot Phase (IIV4) | Study Phase (LAIV4) | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7.93) |  | 32 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0
Population: Study halted after Pilot Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Phase | Study Phase
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

2. Primary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 14 post-immunization
Measure: Count of Participants; unit: Participants
Groups:
- Pilot Phase (IIV4): Participants will receive the current seasonal quadrivalent, inactivated influenza vaccine (IIV4)/Fluzone® given intramuscularly to confirm the safety of administering the seasonal influenza vaccine 3-14 days prior to tonsillectomy.
  Fluzone®: quadrivalent, inactivated influenza virus vaccine, intramuscular
- Study Phase (LAIV4): Participants will be given the current year's quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4)/FluMist® intranasally 3-14 days prior to tonsillectomy.
  FluMist®: quadrivalent, live, attenuated influenza vaccine, intranasal spray
Arm/Group | Pilot Phase (IIV4) | Study Phase (LAIV4)
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Pilot Phase (IIV4) | Study Phase (LAIV4)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No